CLINICAL TRIAL: NCT06061497
Title: Effectiveness of a Rehabilitation Nursing Consultation for People With Asthma
Brief Title: Effectiveness of the Rehabilitation Nursing Consultation for People With Asthma on Symptom Control and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ACES Entre Douro e Vouga II - Aveiro Norte (Other)
Responsible Party: Principal Investigator, Andreia Patrícia de Oliveira Santos, Investigator, ACES Entre Douro e Vouga II - Aveiro Norte
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RehabAsthma
Record Dates: First submitted 2023-09-09; First posted 2023-09-29 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Asthma; Rehabilitation; Breathing, Mouth; Nursing Caries; Adult
Keywords: Asthma; Nurse; Rehabilitation; Quality of life; Breathing exercises; Clinical Trials; Obstructive airway disease; Non-pharmacological therapy
MeSH Terms: conditions — Asthma; Mouth Breathing; Lung Diseases, Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abdomino-diaphragmatic breathing (Experimental): There are four consultations with autonomous rehabilitation nursing intervention: abdomino-diaphragmatic breathing.
  In addition to adding the health care that is recommended in the Integrated Care Process for Asthma in Children and Adults, of the Portuguese Directorate-General for Health, namely:
  Health education:
  Inhalation technique Adherence to treatment; Presence of comorbidities; Smoking; Other environmental factors; Promotion of physical activity.
  Interventions: Other: Abdomino-diaphragmatic breathing; Behavioral: Usual Care
- Usual care (Placebo Comparator): They will have the care recommended in the Integrated Care Process for Asthma in Children and Adults, of the Portuguese Directorate-General for Health, namely:
  Health education:
  Inhalation technique Adherence to treatment; Presence of comorbidities; Smoking; Other environmental factors; Promotion of physical activity.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Other: Abdomino-diaphragmatic breathing — Breathing should be done twice a day for 10 minutes.
  Arms: Abdomino-diaphragmatic breathing
Behavioral: Usual Care — Health education Review of inhaler technique Check adherence to treatment; Presence of comorbidities; Smoking; Other environmental factors; Promotion of physical activity

SUMMARY:
Introduction Asthma is a chronic inflammatory disease of the respiratory airways and is considered a Public Health problem, which lacks a personalized multidisciplinary intervention, to allow the user to develop mastery in the self-management of his disease. The project intends to answer the question: What methods could be used to enhance the use of asthma controller therapy? Methods Randomized and controlled clinical trial. The sample consists of users with asthma at Family Health Units in the municipality of Oliveira de Azeméis. There will be an experimental group that will undergo structured rehabilitation nursing consultations, and a control group that will receive the usual nursing care appropriate for asthma management.

Both groups will be subject to two evaluation moments with the CARAT test and the AQLQ-M questionnaire. Results The aim is to evaluate the effectiveness of interventions for people with asthma implemented within the framework of a structured rehabilitation nursing consultation. The investigators expected to observe a clinically significant improvement with regard to disease control, quality of life, and user empowerment.

DETAILED DESCRIPTION:
By carrying out this study, the following aims are intended to be achieved:

Main Goal To evaluate the effectiveness of rehabilitation nursing interventions in adults with asthma in controlling symptoms and quality of life. Specific Goals To evaluate the symptomatic improvement, comparing the initial and final evaluation.

To evaluate the quality of life related to health, comparing the initial and final evaluation after consultations, using the Asthma Quality Of Life Questionnaire by Marks (AQLQ-M); To achieve the proposed objectives, the investigators started with the following question: What are the effects of a structured rehabilitation nursing consultation on asthma control and healthrelated quality of life? To answer this question, a randomized and controlled clinical trial will be carried out, with the intention of studying the effectiveness of the interventions under study, comparing them with usual care. The population under study are people with asthma, the sample being made up of adults with asthma, enrolled in the ACeS Entre Douro e Vouga II, belonging to the municipality of Oliveira de Azeméis. The sample will be consecutive non-random.

Participants will be randomly assigned to one of 2 groups, intervention or control. The encryption key will be prepared using MS Excel and will be filed in a closed cabinet under the responsibility of the principal investigator. The minimum necessary sample size was calculated considering the final comparison between the two groups. Therefore, stipulating the T test for independent samples as the procedure to be used, or the corresponding non-parametric Mann-Whitney U test, a significance level of 5%, a test power (1-β) of 80%, an effect magnitude high, the sample size to be collected will be 102 participants, which corresponds to 51 participants per group. Considering that the investigators may have 20% of follow-up losses, the sample size to be collected will be 102 participants (51 per group). Participants in both groups will be subject to two evaluation moments, an initial one during the first contact and another at the end of the intervention.

The following variables will be studied:

Independent variable Structured rehabilitation nursing consultation for people with asthma.

Main dependent variable:

* Asthma control - assessed with the Asthma and Allergic Rhinitis Control Test (CARAT) Secondary dependent variables
* Quality of life - assessed with the Asthma-Related Quality of Life Questionnaire (AQLQ - M)
* User empowerment - assessed with mPEI modified Patient Enablement Instrument. Intervention Both groups will have access to the health care recommended in the Integrated Care

Process for Asthma in Children and Adults, of the DGS, namely:

* Education for health;
* Inhalation technique;
* Adherence to treatment;
* Presence of comorbidities;
* Smoking;
* Other environmental factors;
* Promotion of physical activity. The rehabilitation nursing consultation will be carried out by the specialist nurse in rehabilitation nursing, at UCC Aveiro Norte, during the year 2023 and will be based on autonomous interventions in the domain of the specialist nurse in rehabilitation nursing, within the scope of training for self-management of asthma, breathing exercises. These interventions are in addition to those implemented in a Nursing consultation, for the person with asthma defined by the DGS and which will be applied in the control group, first consultation and in the fourth week. The Intervention group will be held during four consultations, one per week, where the following interventions will be carried out:
* Breathing awareness and control;
* Postural correction techniques;
* Relaxation techniques and resting positions;
* Airway permeabilization techniques

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma, with R96 coding according to ICPC2;
* Users enrolled in health units in the municipality of Oliveira de Azeméis.

Exclusion Criteria:

* Impossibility of contacting the user to schedule the appointment;
* Users with severe cognitive dysfunction or psychiatric illness with interference in memory and adherence;
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2023-07-03 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Symptom Control using the scale Allergic Rhinitis and Control of Asthma Test CARAT | At the first and last consultation in 4 weeks
  The CARAT questionnaire is composed of 10 questions that address upper and lower airway symptoms, sleep interference, activity limitation, and the need to increase medication over a four-week period. Scores above 24 indicate good disease control.
  Upper airway score (item 1-4): 0 Controlled if score >8 Lower airway score (item 5-10): 0 Controlled if score ≥16
Quality of life in asthma patients using the scale Mini Ashma Quality of Life Questionnaire (Mini- AQLQ) | At the first and last consultation in 4 weeks
  This instrument has 15 questions in the same domains as the original AQLQ (symptoms, activities, emotions and environment) and takes 3-4 minutes to complete. An increase of 0.5 in the Mini-AQLQ score is considered a clinically significant improvement.
Measure patient enablement in asthma using the scale mPEI | At the last consultation, an average of 4 weeks after the first consultation
  The mPEI is a six-item questionnaire. Each item is scored in a Likert-type scale from 0 ('same or less' or 'not applicable') to 2 ('much better'). There is a minimum score of 0 and a maximum score of 12. A higher score reflects higher patient enablement

CONTACTS AND LOCATIONS:
Overall Officials: Andreia Santos, Principal Investigator — ACES Entre Douro e Vouga II
Locations (1):
- ACES Entre Douro e Vouga II- Aveiro Norte, Oliveira de Azeméis, Aveiro District, Portugal

IPD SHARING:
Plan to Share IPD: No